CLINICAL TRIAL: NCT01878825
Title: Immunogenicity and Safety Study of GSK Biologicals' Trivalent Split Virion Influenza Vaccine (GSK1536489A) Fluviral™ (2013-2014 Season) in Adults Aged 18 Years and Older
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Trivalent Split Virion Influenza Vaccine Fluviral™ (2013-2014 Season) in Adults Aged 18 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200190
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-06

CONDITIONS: Influenza
Keywords: Immunogenicity; Trivalent; Safety; Adults; Elderly; Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

ARMS (2):
- Fluviral 18-60 Years Group (Experimental): Subjects aged between 18 and 60 years, received 1 dose of Fluviral™ vaccine on Day 0. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluviral™
- Fluviral >60 Years Group (Experimental): Subjects aged > 60 years, received 1 dose of Fluviral™ vaccine on Day 0. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm
  Interventions: Biological: Fluviral™

INTERVENTIONS:
Biological: Fluviral™ — 1 dose administered intramuscularly in deltoid region of non-dominant arm.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, reactogenicity and safety of Fluviral™ containing the influenza strains recommended for the 2013-2014 season in adults aged 18 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female 18 years of age and older at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects or subjects with well-controlled chronic disease, as established by medical history and clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination dose.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose. For corticosteroids, this will mean prednisone ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Any administration of a long-acting immune-modifying drug (e.g. rituximab, infliximab etc.) within 6 months before study start, or planned administration during the study period.
* Administration of any influenza vaccine within 6 months preceding the study start or planned use of such vaccines during the study period.
* Administration of any other vaccine(s) within 30 days prior to study enrollment or during the study period.
* Clinically or virologically confirmed influenza infection within the 6 months preceding the study vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required):

  * History of human immunodeficiency virus (HIV) infection,
  * Cancer or treatment for cancer, within 3 years of study enrollment. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* Acute disease and/or fever at the time of enrollment.

  * Acute disease is defined as the presence of a short term, moderate or severe illness, with or without fever.
  * Fever is defined as temperature ≥ 38.0°C/100.4°F for oral, axillary or tympanic route. The preferred route for recording temperature in this study will be oral.
  * Subjects with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Significant acute or chronic, uncontrolled medical or psychiatric or neurological illness. "Uncontrolled" is defined as:

  * Requiring institution of new medical or surgical treatment within one month prior to study enrollment, or
  * Requiring the re-institution of a previously discontinued medication or medical treatment within one month prior to study enrollment, or
  * Requiring a change in medication dosage in the one month prior to study enrollment due to uncontrolled symptoms or drug toxicity (elective dosage adjustments in stable subjects are acceptable), or
  * Hospitalization or an event fulfilling the definition of a SAE within one month prior to study enrollment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Subjects who participated in the registration trial [116664 (FLU Q-TIV-014)] for Fluviral™ 2012/2013 conducted in the 2012-2013 season.
* Presence of blood dyscrasias, including hemoglobinopathies and myelo- or lymphoproliferative disorder.
* A history of any demyelinating disease including Multiple Sclerosis and Guillain-Barré syndrome.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study vaccine or planned administration during the study period.
* Any known or suspected allergy to any constituent of Fluviral™ and/or a history of anaphylactic type reaction to consumption of eggs, and/or reactions to products containing mercury.
* A history of severe adverse reaction to a previous influenza vaccination.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study or would make the intramuscular injection unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-07-18; Primary Completion 2013-08-09 (Actual); Study Completion 2013-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 volunteer was assigned a subject number but was subsequently determined to be ineligible for study participation and was never vaccinated.
Period: Overall Study
Arm/Group | Fluviral 18-60 Years Group | Fluviral >60 Years Group
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluviral 18-60 Years Group | Fluviral >60 Years Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.1 (11.63) | 68.6 (4.92) | 54.9 (16.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 32 | 72
  Male | 20 | 28 | 48

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibody Titers Against Each of the Three Vaccine Influenza Strains
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Days 0 and 21
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Fluviral 18-60 Years Group | Fluviral >60 Years Group
Number analyzed (Participants) | 59 | 60
Titer
  H1N1, Day 0 | 61.0 [41.2 to 90.5] | 65.7 [48.6 to 88.9]
  H1N1, Day 21 | 337.4 [260.9 to 436.3] | 207.5 [163.3 to 263.5]
  H3N2, Day 0 | 37.3 [26.9 to 51.6] | 31.5 [23.3 to 42.7]
  H3N2, Day 21 | 159.0 [124.1 to 203.8] | 133.7 [101.5 to 176.2]
  Yamagata, Day 0 | 200.0 [150.3 to 266.1] | 159.0 [118.0 to 214.3]
  Yamagata, Day 21 | 521.1 [417.9 to 649.8] | 407.8 [328.9 to 505.7]

2. Primary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluviral 18-60 Years Group | Fluviral >60 Years Group
Number analyzed (Participants) | 59 | 60
Subjects
  H1N1 | 32 | 22
  H3N2 | 24 | 25
  Yamagata | 21 | 17

3. Primary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Three Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluviral 18-60 Years Group | Fluviral >60 Years Group
Number analyzed (Participants) | 59 | 60
Fold increase
  H1N1 | 5.5 [3.5 to 8.6] | 3.2 [2.2 to 4.4]
  H3N2 | 4.3 [3.0 to 6.1] | 4.2 [3.0 to 6.0]
  Yamagata | 2.6 [1.9 to 3.5] | 2.6 [1.9 to 3.5]

4. Primary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Days 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluviral 18-60 Years Group | Fluviral >60 Years Group
Number analyzed (Participants) | 59 | 60
Subjects
  H1N1, Day 0 | 41 | 44
  H1N1, Day 21 | 59 | 59
  H3N2, Day 0 | 37 | 33
  H3N2, Day 21 | 56 | 54
  Yamagata, Day 0 | 55 | 56
  Yamagata, Day 21 | 59 | 60

5. Secondary Outcome: Humoral Immune Response in Terms of HI Antibody Titers Against Each of the Three Vaccine Influenza Strains
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata). This outcome measure was assessed by influenza vaccination status in subjects (18-60 years and >60 years) who had and who had not received an influenza vaccine during the 2012/2013 influenza season.
Time Frame: At Days 0 and Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Fluviral 18-60 Years Group With Vaccination: Subjects 18-60 years of age received 1 dose of Fluviral™ 2013-2014 vaccine at Day 0 and who had received an influenza vaccine during the 2012-2013 influenza season. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluviral 18-60 Years Group Without Vaccination: Subjects 18-60 years of age received 1 dose of Fluviral™ 2013-2014 vaccine at Day 0 and who had not received an influenza vaccine during the 2012-2013 influenza season. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluviral >60 Years Group With Vaccination: Subjects above 60 years of age received 1 dose of Fluviral™ 2013-2014 vaccine at Day 0 and who had received an influenza vaccine during the 2012-2013 influenza season. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluviral > 60 Years Group Without Vaccination: Subjects above 60 years of age received 1 dose of Fluviral™ 2013-2014 vaccine at Day 0 and who had not received an influenza vaccine during the 2012-2013 influenza season. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | Fluviral 18-60 Years Group With Vaccination | Fluviral 18-60 Years Group Without Vaccination | Fluviral >60 Years Group With Vaccination | Fluviral > 60 Years Group Without Vaccination
Number analyzed (Participants) | 29 | 30 | 30 | 30
Titers
  H1N1, Day 0 | 132.2 [91.6 to 190.8] | 28.9 [16.0 to 52.2] | 70.5 [49.2 to 100.9] | 61.3 [36.9 to 101.8]
  H1N1, Day 21 | 249.0 [177.6 to 349.0] | 452.6 [311.4 to 657.7] | 136.1 [105.1 to 176.2] | 316.3 [222.0 to 450.7]
  H3N2, Day 0 | 58.6 [38.1 to 90.2] | 24.1 [15.3 to 38.0] | 47.5 [32.5 to 69.6] | 20.9 [13.4 to 32.7]
  H3N2, Day 21 | 107.9 [78.1 to 148.9] | 231.5 [165.1 to 324.6] | 109.3 [75.8 to 157.4] | 163.6 [107.3 to 249.5]
  Yamagata, Day 0 | 352.1 [250.2 to 495.4] | 115.8 [79.8 to 168.0] | 218.6 [160.0 to 298.6] | 115.7 [70.1 to 191.1]
  Yamagata, Day 21 | 436.7 [319.0 to 597.6] | 618.2 [450.8 to 847.8] | 342.9 [259.9 to 452.3] | 485.0 [347.4 to 677.1]

6. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata).This outcome measure was assessed by influenza vaccination status in subjects (18-60 years and >60 years) who had and who had not received an influenza vaccine during the 2012/2013 influenza season.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Groups:
- Fluviral > 60 Years Group With Vaccination: Subjects above 60 years of age received 1 dose of Fluviral™ 2013-2014 vaccine at Day 0 and who had received an influenza vaccine during the 2012-2013 influenza season. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
- Fluviral >60 Years Group Without Vaccination: Subjects above 60 years of age received 1 dose of Fluviral™ 2013-2014 vaccine at Day 0 and who had not received an influenza vaccine during the 2012-2013 influenza season. The vaccine was administered intramuscularly in the deltoid of the non-dominant arm.
Arm/Group | Fluviral 18-60 Years Group With Vaccination | Fluviral 18-60 Years Group Without Vaccination | Fluviral > 60 Years Group With Vaccination | Fluviral >60 Years Group Without Vaccination
Number analyzed (Participants) | 29 | 30 | 30 | 30
Subjects
  H1N1 | 7 | 25 | 6 | 16
  H3N2 | 4 | 20 | 7 | 18
  Yamagata | 2 | 19 | 3 | 14

7. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Three Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata). This outcome measure was assessed by influenza vaccination status in subjects (18-60 years and >60 years) who had and who had not received an influenza vaccine during the 2012/2013 influenza season.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluviral 18-60 Years Group With Vaccination | Fluviral 18-60 Years Group Without Vaccination | Fluviral > 60 Years Group With Vaccination | Fluviral > 60 Years Group Without Vaccination
Number analyzed (Participants) | 29 | 30 | 30 | 30
Fold increase
  H1N1 | 1.9 [1.4 to 2.5] | 15.6 [8.2 to 29.9] | 1.9 [1.5 to 2.5] | 5.2 [2.9 to 9.3]
  H3N2 | 1.8 [1.4 to 2.4] | 9.6 [5.7 to 16.1] | 2.3 [1.6 to 3.2] | 7.8 [4.5 to 13.6]
  Yamagata | 1.2 [1.0 to 1.5] | 5.3 [3.5 to 8.1] | 1.6 [1.3 to 1.9] | 4.2 [2.5 to 7.1]

8. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against Each of the Three Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2) and Flu B/Massachusetts/2/2012 (Yamagata). This outcome measure was assessed by influenza vaccination status in subjects (18-60 years and >60 years) who had and who had not received an influenza vaccine during the 2012/2013 influenza season.
Time Frame: At Day 0 and Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluviral 18-60 Years Group With Vaccination | Fluviral 18-60 Years Group Without Vaccination | Fluviral >60 Years Group With Vaccination | Fluviral > 60 Years Group Without Vaccination
Number analyzed (Participants) | 29 | 30 | 30 | 30
Subjects
  H1N1, Day 0 | 27 | 14 | 23 | 21
  H1N1, Day 21 | 29 | 30 | 29 | 30
  H3N2, Day 0 | 22 | 15 | 20 | 13
  H3N2, Day 21 | 27 | 29 | 26 | 28
  Yamagata, Day 0 | 29 | 26 | 30 | 26
  Yamagata, Day 21 | 29 | 30 | 30 | 30

9. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were ecchymosis, induration, pain, redness and swelling. Any was defined as any solicited local symptom reported irrespective of intensity. Grade 3 pain was defined as pain that prevented normal everyday activities. Grade 3 ecchymosis, induration, redness and swelling was greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: Analysis was performed on the Total Vaccinated cohort, which included all subjects with vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Fluviral 18-60 Years Group | Fluviral >60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects
  Any Ecchymosis | 0 | 0
  Grade 3 Ecchymosis | 0 | 0
  Any Induration | 2 | 1
  Grade 3 Induration | 0 | 0
  Any Pain | 42 | 15
  Grade 3 Pain | 0 | 0
  Any Redness | 0 | 0
  Grade 3 Redness | 0 | 0
  Any Swelling | 5 | 2
  Grade 3 Swelling | 0 | 0

10. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering, increased sweating and fever [oral temperature above 37.5 degrees Celsius (°C)]. Gastrointestinal symptoms included nausea, vomiting, diarrhea and/or abdominal pain. Any = any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related = symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 fever = oral temperature above 39.0°C
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 9
Measure: Number; unit: Subjects
Groups:
- Fluarix/Influsplit 18-60 Years Group: Subjects aged between 18 and 60 years, received 1 dose of Fluviral™ vaccine on Day 0. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm
- Fluarix/Influsplit > 60 Years Group: Subjects aged > 60 years, received 1 dose of Fluviral™ vaccine on Day 0. The vaccine was administered intramuscularly in the deltoid region of the non-dominant arm
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects
  Any Arthralgia | 4 | 5
  Grade 3 Arthralgia | 0 | 1
  Related Arthralgia | 4 | 5
  Any Fatigue | 9 | 6
  Grade 3 Fatigue | 0 | 1
  Related Fatigue | 9 | 6
  Any Gastrointestinal symptoms | 4 | 3
  Grade 3 Gastrointestinal symptoms | 0 | 1
  Related Gastrointestinal symptoms | 4 | 3
  Any Headache | 6 | 6
  Grade 3 Headache | 0 | 2
  Related Headache | 6 | 6
  Any Myalgia | 18 | 6
  Grade 3 Myalgia | 0 | 1
  Related Myalgia | 18 | 6
  Any Shivering | 0 | 1
  Grade 3 Shivering | 0 | 0
  Related Shivering | 0 | 1
  Any Sweating | 0 | 3
  Grade 3 Sweating | 0 | 1
  Related Sweating | 0 | 3
  Any Fever ( ≥ 37.5°C) | 2 | 1
  Grade 3 Fever (>39.0°C) | 0 | 0
  Related Fever | 2 | 1

11. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 21-day (Days 0-20) post-vaccination period
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects | 9 | 7

12. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: A serious adverse event was any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (Days 0-20 post vaccination)
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Number analyzed (Participants) | 60 | 60
Subjects | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 20 post vaccination; Solicited local and general symptoms: During the 4-day (Days 0-3) post-vaccination period; Unsolicited symptoms: During the 21-day (Day 0-20) post-vaccination period
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | Fluarix/Influsplit 18-60 Years Group | Fluarix/Influsplit > 60 Years Group
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 45/60 | 23/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix/Influsplit 18-60 Years Group (N=60) | Fluarix/Influsplit > 60 Years Group (N=60)
Pain (General disorders) | 42 | 15
Swelling (General disorders) | 5 | 2
Arthralgia (General disorders) | 4 | 5
Gastrointestinal symptoms (General disorders) | 4 | 3
Headache (General disorders) | 6 | 6
Myalgia (General disorders) | 18 | 6
Sweating (General disorders) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Fatigue (General disorders) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.